CLINICAL TRIAL: NCT01632449
Title: A Randomized, Single-Blind, Two-Period Crossover Study in Healthy Volunteers to Establish the Bioequivalence of BG00012 Supplied by Two Different Manufacturers.
Brief Title: Study in Healthy Volunteers to Establish the Bioequivalence of Two Different Manufacturers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 109HV109
Record Dates: First submitted 2012-06-21; First posted 2012-07-03 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Volunteers
Keywords: bioequivalence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Test product
  Interventions: Drug: Test product; Drug: Reference product
- 2 (Experimental): Reference product
  Interventions: Drug: Test product; Drug: Reference product

INTERVENTIONS:
Drug: Test product — Dimethyl Fumarate (BG00012)
Drug: Reference product — Dimethyl Fumarate (BG00012)

SUMMARY:
This is an single-blind, single-center, two-period crossover, PK profile study. Each subject will be randomized to one of two treatment sequences. Both treatment sequences will be enrolled concurrently.

DETAILED DESCRIPTION:
This is a study of healthy volunteers to demonstrate bioequivalence of one formulation of BG-00012 given in capsule form supplied by two different manufactures.

ELIGIBILITY:
Inclusion Criteria:

* Must give written and informed consent and any authorizations required by local law.
* Males and females 18 - 55 years old inclusive at time of consent.
* Must have a body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive

Exclusion Criteria:

* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic,metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric and renal or other major disease, as determined by the Investigator.
* Clinically significant abnormal hematology or blood chemistry values, as determined by the Investigator, and any screening values for alanine aminotransferase (ALT) aspartate aminotransferase (AST) total bilirubin, or creatinine above the upper limit of normal, or an out of normal range screening value for white blood cells (WBC).
* Current enrollment in any other drug, biologic, or device study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
PK - Area under the plasma concentration curve. | Participants will be followed during the duration of the study, 4 days. Thirteen samples taken over the course of approximately 12 hours
Peak plasma concentration as a measure of PK. | Participants will be followed during the duration of the study, 4 days. Thirteen samples taken over the course of approximately 12 hours

SECONDARY OUTCOMES:
The number of AEs in participants as a measure of safety and tolerability. | Participants will be followed during the study, 4 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Minneapolis, Minnesota, United States